CLINICAL TRIAL: NCT00173147
Title: Morphology of the Vastus Medialis Obliquus in Patients With Patellofemoral Pain Syndrome and Healthy Young Adults --A Sonographic Study
Brief Title: Morphology of the VMO in Patients With PFPS and Healthy Young Adults--A Sonographic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700502
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2005-04

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background：Patellofemoral pain syndrome（PFPS） is a common knee disorder characterized by anterior or retropatellar pain associated with activities that load the patellofemoral joint. Previous studies reveal that the vastus medialis obliquus（VMO） is an important dynamic medial stabilizer of the patellar. Insufficiency of the VMO leads to lateral shift of the patella and the increases the patellofemoral contact force. An in vitro study conducted by Hubbard JK. et al. claimed that there were no significant relationship between several morphologic characteristics of the VMO and the extent of patellofemoral joint deterioration. We consider that the condition might be different in vivo, so we chose ultrasonogrphy as the measurement tool to examine the morphology of the VMO in PFPS patients and healthy controls. Purpose：To determine if there are significant differences in several morphologic parameters of the VMO between patients with PFPS and healthy controls under 50. Method：31 PFPS patients and 31 matched healthy adults under 50 were recruited for the study. The HDI 5000 ultrasonography machine was used to evaluate morphologic parameters of the VMO, including the percent of patella attachment, fiber angle, the volume attached to the patella, and the change of shape of the VMO.

ELIGIBILITY:
Inclusion Criteria:

1. under 50 years old.
2. Have a diagnosis of PFPS.

Exclusion Criteria:

1. Diagnosis other than PFPS，such as meniscal lesion, ligamentous instability ,patellar tendon pathology, traction apophysitis, radiation pain, referred pain, ect.
2. Knee operation within three month.
3. X-ray findings (1)joint space narrowing (2)osteophyte formation

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwa Jan, Master, Study Chair — NTU department of physical therapy
Locations (1):
- NTUH, Taipei, Taiwan